CLINICAL TRIAL: NCT00002408
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Orally Administered SP-303 for the Treatment of Diarrhea in Acquired Immunodeficiency Syndrome (AIDS) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaman Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 293A; 37,554-210
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: Diarrhea; HIV Infections
Keywords: Diarrhea; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Diarrhea; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — crofelemer

INTERVENTIONS:
Drug: Crofelemer

SUMMARY:
To evaluate the efficacy, safety, and durability of response of SP-303 in decreasing stool weight in AIDS patients with diarrhea over 6 days of treatment.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection meeting CDC criteria for AIDS.
* History of diarrhea for greater than or equal to 14 days prior to screening period (Day 1).

Required:

- On stable medical regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (36):
- United States (34):
  - Hill Top Research Ltd, Scottsdale, Arizona
  - Phoenix Living Ctr, Scottsdale, Arizona
  - UCLA Care Ctr, Los Angeles, California
  - AIDS Research Ctr / Dept of Veterans Affairs, Palo Alto, California
  - San Francisco Gen Hosp, San Francisco, California
  - Lynn House Hospice, West Hollywood, California
  - AIDS Research Alliance, West Hollywood, California
  - Howard Univ, Washington D.C., District of Columbia
  - GCRC, Washington D.C., District of Columbia
  - Community CRI of South Florida, Coral Gables, Florida
  - Central Florida Research Initiative, Maitland, Florida
  - Deering Hosp, Miami, Florida
  - Rosemont Health Care Ctr, Orlando, Florida
  - Ctr for Quality Care, Tampa, Florida
  - Mem Hosp of Tampa, Tampa, Florida
  - Phillip Branchman, Atlanta, Georgia
  - Insite Clinical Trials, Decatur, Georgia
  - Oak Park Hosp, Oak Park, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - New Orleans Pharmaceutical Research, Kenner, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Wayne State Univ, Detroit, Michigan
  - Hennepin County Med Ctr, Minneapolis, Minnesota
  - Regions Hosp, Saint Paul, Minnesota
  - Washington Univ School of Medicine, St Louis, Missouri
  - Brookdale Univ Hosp and Med Ctr, Brooklyn, New York
  - Saint Vincents Hosp, New York, New York
  - Wake Med CRI, Raleigh, North Carolina
  - Joseph Gathe, Houston, Texas
  - GCRC - VA Hosp, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Bailey Boushay House, Seattle, Washington
  - Rosehedge House, Seattle, Washington
- Puerto Rico (2):
  - Hosp Regional de Ponce, Ponce
  - Clinical Research Puerto Rico Inc, San Juan